CLINICAL TRIAL: NCT07368452
Title: Video-Based Versus Simulation-Based Basic Life Support Training in Medical Students: A Randomized Trial
Brief Title: Video-Based Versus Simulation-Based Basic Life Support Training in Medical Students
Acronym: BLS-VIDEO-SIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Serkan TELLİ, Assistant Proffesor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/11-45
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Medical Education; Cardiopulmonary Resuscitation (CPR); Basic Life Support (BLS) Training
Keywords: basic life support; cardiopulmonary resuscitation; simulation-based education; video-based education; OSCE

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two parallel arms (video-based vs simulation-based BLS training) and received only the assigned intervention.
Who Masked: Outcomes Assessor
Masking Description: Masking Description: Not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based BLS training (Experimental): Participants received a structured video-based Basic Life Support (BLS) training module covering adult CPR and AED use, delivered as standardized instructional videos. After viewing the module, participants completed the planned practice session(s) according to the curriculum and subsequently underwent the scheduled assessments.
  Interventions: Behavioral: Video-based BLS training
- Simulation-based BLS training (Experimental): Participants received instructor-led, simulation-based Basic Life Support (BLS) training using manikins and scenario-based practice focused on adult CPR and AED use. Training was delivered according to the curriculum, followed by the scheduled assessments.
  Interventions: Behavioral: Simulation-based BLS training

INTERVENTIONS:
Behavioral: Video-based BLS training — A structured video-based Basic Life Support (BLS) training module covering adult CPR and AED use, delivered via standardized instructional videos.
  Arms: Video-based BLS training
Behavioral: Simulation-based BLS training — Instructor-led simulation-based Basic Life Support (BLS) training using manikins and scenario-based practice focused on adult CPR and AED use.
  Arms: Simulation-based BLS training

SUMMARY:
This randomized educational trial compared a structured video-based Basic Life Support (BLS) training program with simulation-based BLS training among fourth-year medical students. Participants were allocated to one of the two training formats and completed a BLS knowledge test before and immediately after training. Performance was assessed using an Objective Structured Clinical Examination (OSCE) conducted 3 weeks after training. The primary outcome was OSCE performance at 3 weeks, and secondary outcomes included knowledge test scores and knowledge gain.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment as a fourth-year medical student at the study institution
* Age 18 years or older
* Willingness to participate in the study
* Provision of written informed consent

Exclusion Criteria:

* Previous participation in a formal BLS instructor or trainer program
* Declined or withdrew informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2025-10-04 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
OSCE performance score | 3 weeks after training
  Total score obtained on a standardized Basic Life Support (BLS) Objective Structured Clinical Examination (OSCE) checklist. Higher scores indicate better performance.

SECONDARY OUTCOMES:
BLS knowledge test score (pre-test) | Baseline (before training)
  Score obtained on a multiple-choice BLS knowledge test administered before training.
BLS knowledge test score (post-test) | Immediately after training
  Score obtained on the same multiple-choice BLS knowledge test administered immediately after training.

OTHER OUTCOMES:
Knowledge gain | From baseline to immediately after training
  Change in BLS knowledge test score calculated as post-test score minus pre-test score.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly, as the dataset contains institution-specific educational assessment data and sharing was not included in the original ethics approval. De-identified aggregate data are reported in the manuscript.